CLINICAL TRIAL: NCT00438113
Title: Atrial Substrate Modification With Aggressive Blood Pressure Lowering to Prevent AF
Acronym: SMAC AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Principal Investigator, Ratika Parkash, Staff Cardiologist, Electrophysiology, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RP-001
Record Dates: First submitted 2007-02-07; First posted 2007-02-21 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Atrial Fibrillation
Keywords: blood pressure; atrial fibrillation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Quinapril; Atenolol; Amlodipine; Terazosin; Hydrochlorothiazide

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aggressive Blood Pressure control (Active Comparator): The experimental arm will receive open label therapy to achieve a target systolic blood pressure less than or equal to 120 mmHg.
  If the average BP is found to be > 120 mmHg at the baseline, telephone or clinic followup visits, treatment will be recommended based on the following regimen (For details, please see Appendix 4):
  Step 1 - Accupril, titrated to maximum tolerated dose, beginning at 20 mg po od followed by 40 mg successively Step 2 - combination of Accupril with Hydrochlorothiazide 12.5 mg po od. Step 3 - Addition of Atenolol 50 mg po od. Step 4 - Addition of Norvasc 2.5-10 mg po od. Step 5 - Addition of Terazosin 1 mg po od.
  Interventions: Drug: Aggressive Blood Pressure control
- Standard Blood Pressure control (No Intervention): Treatment will be carried out as per the CHEP guidelines. These patients may require ACEi or ARBs for their treatment. No changes to their drug regimen will be made as long as BP measurements are congruent with current guidelines. These modifications will be made as per standard practice by the physician who is primarily involved with their care (this may be a family physician or a specialist, depending on the patient). Patients with diabetes in the standard arm will be treated to a target BP of <130/80 as per the CHEP guidelines.

INTERVENTIONS:
Drug: Aggressive Blood Pressure control — Aggressive Blood Pressure therapy, alone or combination therapy, to reach a target BP equal to or less than 120/80 mmHg
  Other Names: Accupril; Atenolol; Norvasc; Terazosin; Hydrochlorothiazide
  Arms: Aggressive Blood Pressure control

SUMMARY:
Atrial fibrillation (AF) is a very common arrhythmia causing many symptoms resulting in numerous hospitalizations. Catheter ablation is a technique that has evolved significantly to improve symptomatic recurrences, but does not offer a 100% cure rate. We hypothesize that the use of aggressive BP lowering will reduce the rate of recurrent AF after catheter ablation for AF. We plan a randomized clinical trial of aggressive BP lowering versus standard BP control to investigate this.

DETAILED DESCRIPTION:
Background: Atrial fibrillation (AF) is the most common sustained arrhythmia and is associated with significant morbidity, necessitating treatment. Radiofrequency ablation for atrial fibrillation/flutter has evolved significantly and is the closest we have come to a 'cure' for these dysrhythmias. Recurrence of atrial fibrillation in those who have undergone radiofrequency ablation as treatment AF is up to 40% at one year and higher in those with persistent AF. Hypertension is a potent risk factor for AF, but recent studies have demonstrated that even modest increases in BP may lead to a higher incidence of AF. There is no clinical trial evidence to date that has investigated aggressive BP control in patients post radiofrequency ablation for AF to prevent recurrent AF.

Objective: We propose to determine if aggressive BP control reduces recurrent AF post ablation.

Hypothesis: Aggressive BP lowering will reduce the incidence of recurrent AF post ablation.

Research Plan:

Study Design. This will be a randomized open label trial in patients who are post catheter ablation for atrial fibrillation. Randomization to either aggressive BP lowering or standard BP control will occur three to six months prior to the procedure.

Study Population. Patients will be included if they have persistent or high burden paroxysmal (refractory to class 1 or 3 antiarrhythmic medication) and intend to have a catheter ablation procedure for AF.

Followup. Patients will be followed at 3 month intervals for the first year, then every 6 months to a maximum of 30 months or the common study end date has been reached (1 year post randomization for the last patient enrolled).

Statistical Analysis. Kaplan-Meier analysis of the primary outcome will be performed. A Cox proportional hazards model will be constructed to assess the effect of variables chosen a priori on the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Documented systolic blood pressure greater than or equal to 130 mmHg
* Undergoing planned catheter ablation for persistent AF (lasting > 7 days and < 365 days or requiring electrical or chemical cardioversion) OR High burden paroxysmal AF > 6 months (greater than or equal to 3 symptomatic episdes in past 6 months and refractory or inteolerant to at least 1 class 1 or 3 antiarrhythmic)

Exclusion Criteria:

* Permanent atrial fibrillation
* Contraindication to Accupril or any other ACE-I
* Women of child-bearing potential
* Life expectancy less than 1 year
* Less than 18 years of age
* Unable to give informed consent
* Known moderate to several renal dysfunction (eGFR < 30 ml/min/1.73m2)
* Prior AF catheter ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to symptomatic AF/atrial tachycardia (AT)/atrial flutter (AFl) lasting > 30 seconds more than 3 months post ablation. | at least 3 months post catheter ablation
  This has been altered since the inception of the study to include atrial tachycardia and atrial flutter, as there have been changes to how ablation is performed since the study began. Specifically, the STAR AF2 study found that PVI is similar to PVI in addition to either complex fractionated electrogram ablation or PVI in addition to linear ablation. Given this, the occurrence of AT/AFL was thought to be iatrogenic and occur as a consequence of various ablation strategies, rather than to the substrate, hence was excluded from the primary endpoint. Given the change in strategy of ablation, the inclusion of AT/AFl in the primary outcome is now necessary as it may reflect change in substrate, rather than ablation strategy, as previously thought. In addition, from a patient perspective, the occurence of AT/AFl is indistinguishable from a symptoms point of view.

SECONDARY OUTCOMES:
Any recurrent atrial fibrillation/atrial tachycardia/atrial flutter post randomization | up to 30 months post randomization
Recurrent atrial fibrillation/atrial tachycardia/atrial flutter (symptomatic or asymptomatic) post ablation | up to 30 months post randomization
atrial fibrillation/atrial tachycardia/atrial flutter burden (pre and post ablation) | up to 30 months post randomization
Generic and disease specific quality of life | 12 months
Correlation of BNP and CRP and recurrence of atrial fibrillation/atrial tachycardia/atrial flutter | 12 months
Recurrent AF ablation therapy | up to 30 months post randomization
Visits to the ER or hospitalization for atrial arrhythmia | up to 30 months post randomization
Thromboembolic events | up to 30 months post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ratika Parkash, MD MSc, Principal Investigator — Dalhousie University/QEII HSC
Locations (1):
- QE II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weng W, Choudhury R, Sapp J, Tang A, Healey JS, Nault I, Rivard L, Greiss I, Bernick J, Parkash R. The role of brain natriuretic peptide in atrial fibrillation: a substudy of the Substrate Modification with Aggressive Blood Pressure Control for Atrial Fibrillation (SMAC-AF) trial. BMC Cardiovasc Disord. 2021 Sep 16;21(1):445. doi: 10.1186/s12872-021-02254-5. PMID 34530738
- [Derived] Parkash R, Wells GA, Sapp JL, Healey JS, Tardif JC, Greiss I, Rivard L, Roux JF, Gula L, Nault I, Novak P, Birnie D, Ha A, Wilton SB, Mangat I, Gray C, Gardner M, Tang ASL. Effect of Aggressive Blood Pressure Control on the Recurrence of Atrial Fibrillation After Catheter Ablation: A Randomized, Open-Label Clinical Trial (SMAC-AF [Substrate Modification With Aggressive Blood Pressure Control]). Circulation. 2017 May 9;135(19):1788-1798. doi: 10.1161/CIRCULATIONAHA.116.026230. Epub 2017 Feb 22. PMID 28228428